CLINICAL TRIAL: NCT06577142
Title: Comparison of 'Burn 2 Learn' and Routine Physical Activity Program on Wellbeing, Cardiorespiratory and Muscular Fitness Among Students
Brief Title: Burn 2 Learn and Routine Physical Activity Program Among Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0497
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Sports Physical Therapy
Keywords: Exercise; Adolescent health; Cardio-respiratory fitness; High intensity interval training
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 51 participants will be in experimental group giving them ''Burn 2 Learn'' program consisted of high intensity interval training activities such as lunges, jumping jacks, boxing, dancing and sports activities for ten weeks, measuring all values before giving them protocol and after protocol.
  Interventions: Other: Burn 2 Learn
- Group B (Experimental): 51 participants will be in control group participating in their routine school physical activities, sports games or any exercise routines for ten weeks, measuring all values before giving them protocol and after protocol.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Burn 2 Learn — The 'Burn 2 Learn' group encompassed the following components and implementations. A brief introductory seminar will be conducted with the principle, school event coordinator, school sports teacher and students from grade 8 to 10. The aim of this seminar is to provide a better understanding of the rationale and presenting evidence of the beneficial effects of high intensity interval training on overall wellbeing of students. The sessions will be conducted thrice a week for 10 to 15 minutes by the research team members for a period of 10 weeks. The sessions will consist of high intensity interval training activities such as lunges, jumping jacks, boxing, dancing and sports activities. The intervals ranging between 8-16, 30 second work out followed by 30 seconds rest, maintaining a 1:1 work rest ratio.
  51 participants will be in the experimental group A giving them Burn 2 Learn exercise protocol along with the normal sports training plan for ten weeks.
  Arms: Group A
Other: Control Group — 51 participants will be in control group B and will perform their routine school physical activities, sports games or any exercise routines.
  Arms: Group B

SUMMARY:
Engaging in physical activity holds significant benefits for adolescents and contribute to their overall health and well-being. Unfortunately, the younger generation often does not prioritize this aspect of their lifestyle. Schools offer and ideal platform to actively involve and encourage our youth in regular physical activities.

A total of 102 students will be selected from Beaconhouse International School Lahore, who will be passed through screening to fulfill the demands of the inclusion criteria. After selecting students will be randomly assigned into two groups, Group A the 'Burn 2 Learn' group (n=51) and Group B routine physical activity group (n=51). Students in the 'Burn 2 Learn' group will participate in three sessions per week of maximum 20 minutes for 10 weeks. In contrast, students in the routine physical activity group will continue with their routine physical activity implemented within the school. Evaluations of cardiorespiratory fitness using the 20m shuttle run test, wellbeing using the Warwick Edinburgh Mental Wellbeing Scale and muscular fitness using the 90-degree pushup test and standing long jump test, will be taken at baseline and after 10 weeks

DETAILED DESCRIPTION:
The 'Burn 2 Learn' program is a novel approach that integrates physical activity with cognitive engagement in a structured curriculum. The aim of this randomized control trial is to compare the 'Burn 2 Learn' program with routine physical activity on student's cardiorespiratory fitness, wellbeing and muscular fitness.

ELIGIBILITY:
Inclusion Criteria:

* Students aged between 13-16 years (24)
* Students form Grades 8 to 10
* Both male and female students (24)
* Healthy individuals (BMI:18.5 and 24.9) (20)
* Students involved in mild physical activity
* Having playgrounds in school

Exclusion Criteria:

* Students who are differently abled
* Sports injuries
* Students with co morbidities (diabetes)
* Connective tissue disorders
* Mentally retarded students
* Any injury in the upper or lower limb region in the past two years
* Neurological and musculoskeletal disorders that limit movement, and pain in the lower limb prior to and after the tests

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
20-meter Shuttle Run Test | 10 weeks
  The 20- meter shuttle run test, also known as the "Yo-Yo test" or the "Beep test", is a commonly used test for aerobic fitness. It evaluates an individual's aerobic capacity and cardiovascular endurance. The test involves running between two lines that are 20 meters apart in response to audio cues. The speed of the running increases gradually as the speed of the audio beeps increase. The participant must reach the finish line before the beep sounds. The time between beeps gradually decreases and hence the participant increases speed accordingly. If the participant fails to reach the line before the beep, the participant is given a warning. On a second warning, the test is concluded, and the numbers of laps are recorded.
Standing Long Jump Test: | 10 weeks
  The standing long jump test also known as the broad jump test is a commonly used test for lower limb power and strength. It is commonly used in physical education or sports training to check for lower body fitness as it is feasible to perform and does not require much equipment. The test starts with the participant standing at the designated starting line with feet shoulder width apart. The participant then jumps as far as he can from the starting line without any initial run up or step. The distance between the starting lie and the back of the heels where the participant landed is then recorded. After a short interval of rest, the participant is asked to jump again. The best of the two jumps is then recorded.
90 Degree Push Up Test: | 10 weeks
  This test is used to evaluate upper body power and strength, particularly in the chest, shoulders and triceps. The participant assumes a prone position placing hands beneath or slightly wider than the shoulders. The student then lowers the body using the arms until the elbow reaches a 90-degree angle. It is crucial to keep the back in a straight line from head to toe throughout the test. This sequence is repeated as many times as possible in the same form and position. The recommended rhythm is 20 pushups per minute. The test is concluded with a second form correction and the number of pushups is recorded.
Warwick Edinburgh Mental Wellbeing Scale: | 10 weeks
  The Warwick Edinburgh Mental Wellbeing Scale (WEMWBS) is a self-reporting questionnaire consisting of 14 questions designed to assess and individual's mental wellbeing. Data for this questionnaire is gathered through a paper survey filled by the students. Each question is a 5-point scale ranging for "none of the time" to "all the time". The data is filled based on previous two weeks. The items on the Warwick Edinburgh Mental Wellbeing Scale cover areas such as optimism, vitality, relaxation, self-esteem, relationships and overall life satisfaction. The scores from the scale provide a quantitative measure of an individual's mental wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hashim, Principal Investigator — Riphah International University
Locations (1):
- Beaconhouse School Johar Town, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katzmarzyk PT. Expanding our understanding of the global impact of physical inactivity. Lancet Glob Health. 2023 Jan;11(1):e2-e3. doi: 10.1016/S2214-109X(22)00482-X. Epub 2022 Dec 5. No abstract available. PMID 36480932
- [Background] Burden SJ, Weedon BD, Turner A, Whaymand L, Meaney A, Dawes H, Jones A. Intensity and Duration of Physical Activity and Cardiorespiratory Fitness. Pediatrics. 2022 Jul 1;150(1):e2021056003. doi: 10.1542/peds.2021-056003. PMID 35694877
- [Background] Spiga F, Tomlinson E, Davies AL, Moore TH, Dawson S, Breheny K, Savovic J, Hodder RK, Wolfenden L, Higgins JP, Summerbell CD. Interventions to prevent obesity in children aged 12 to 18 years old. Cochrane Database Syst Rev. 2024 May 20;5(5):CD015330. doi: 10.1002/14651858.CD015330.pub2. PMID 38763518
- [Background] Palacios-Cartagena RP, Parraca JA, Mendoza-Munoz M, Pastor-Cisneros R, Munoz-Bermejo L, Adsuar JC. Level of Physical Activity and Its Relationship to Self-Perceived Physical Fitness in Peruvian Adolescents. Int J Environ Res Public Health. 2022 Jan 21;19(3):1182. doi: 10.3390/ijerph19031182. PMID 35162206
- [Background] Cleven L, Krell-Roesch J, Nigg CR, Woll A. The association between physical activity with incident obesity, coronary heart disease, diabetes and hypertension in adults: a systematic review of longitudinal studies published after 2012. BMC Public Health. 2020 May 19;20(1):726. doi: 10.1186/s12889-020-08715-4. PMID 32429951
- [Background] van Sluijs EMF, Ekelund U, Crochemore-Silva I, Guthold R, Ha A, Lubans D, Oyeyemi AL, Ding D, Katzmarzyk PT. Physical activity behaviours in adolescence: current evidence and opportunities for intervention. Lancet. 2021 Jul 31;398(10298):429-442. doi: 10.1016/S0140-6736(21)01259-9. Epub 2021 Jul 21. PMID 34302767
- [Background] Chaput JP, Willumsen J, Bull F, Chou R, Ekelund U, Firth J, Jago R, Ortega FB, Katzmarzyk PT. 2020 WHO guidelines on physical activity and sedentary behaviour for children and adolescents aged 5-17 years: summary of the evidence. Int J Behav Nutr Phys Act. 2020 Nov 26;17(1):141. doi: 10.1186/s12966-020-01037-z. PMID 33239009
- [Background] Zheng W, Shen H, Belhaidas MB, Zhao Y, Wang L, Yan J. The Relationship between Physical Fitness and Perceived Well-Being, Motivation, and Enjoyment in Chinese Adolescents during Physical Education: A Preliminary Cross-Sectional Study. Children (Basel). 2023 Jan 5;10(1):111. doi: 10.3390/children10010111. PMID 36670661
- [Background] Raghuveer G, Hartz J, Lubans DR, Takken T, Wiltz JL, Mietus-Snyder M, Perak AM, Baker-Smith C, Pietris N, Edwards NM; American Heart Association Young Hearts Athero, Hypertension and Obesity in the Young Committee of the Council on Lifelong Congenital Heart Disease and Heart Health in the Young. Cardiorespiratory Fitness in Youth: An Important Marker of Health: A Scientific Statement From the American Heart Association. Circulation. 2020 Aug 18;142(7):e101-e118. doi: 10.1161/CIR.0000000000000866. Epub 2020 Jul 20. PMID 32686505
- [Background] Camacho-Cardenosa A, Amaro-Gahete FJ, Martinez-Tellez B, Alcantara JMA, Ortega FB, Ruiz JR. Sex-specific dose-response effects of a 24-week supervised concurrent exercise intervention on cardiorespiratory fitness and muscular strength in young adults: The ACTIBATE randomized controlled trial. Scand J Med Sci Sports. 2024 Jan;34(1):e14507. doi: 10.1111/sms.14507. Epub 2023 Oct 3. PMID 37787096
- [Background] Barbosa CCL, da Costa JC, Romanzini CLP, Batista MB, Blasquez-Shigaki G, Fernandes RA, Martinho DV, Oliveira T, Ribeiro LP, Coelho-E-Silva MJ, Ronque ERV. Interrelationship between muscle fitness in childhood and bone mineral density in adulthood: mediation analysis of muscle fitness in adulthood. BMC Public Health. 2023 Apr 4;23(1):648. doi: 10.1186/s12889-023-15545-7. PMID 37016376
- [Background] Liu T, Li D, Yang H, Chi X, Yan J. Associations of sport participation with subjective well-being: a study consisting of a sample of Chinese school-attending students. Front Public Health. 2023 Jun 23;11:1199782. doi: 10.3389/fpubh.2023.1199782. eCollection 2023. PMID 37427269
- [Background] Wilhite K, Booker B, Huang BH, Antczak D, Corbett L, Parker P, Noetel M, Rissel C, Lonsdale C, Del Pozo Cruz B, Sanders T. Combinations of Physical Activity, Sedentary Behavior, and Sleep Duration and Their Associations With Physical, Psychological, and Educational Outcomes in Children and Adolescents: A Systematic Review. Am J Epidemiol. 2023 Apr 6;192(4):665-679. doi: 10.1093/aje/kwac212. PMID 36516992
- [Background] Singh AS, Saliasi E, van den Berg V, Uijtdewilligen L, de Groot RHM, Jolles J, Andersen LB, Bailey R, Chang YK, Diamond A, Ericsson I, Etnier JL, Fedewa AL, Hillman CH, McMorris T, Pesce C, Puhse U, Tomporowski PD, Chinapaw MJM. Effects of physical activity interventions on cognitive and academic performance in children and adolescents: a novel combination of a systematic review and recommendations from an expert panel. Br J Sports Med. 2019 May;53(10):640-647. doi: 10.1136/bjsports-2017-098136. Epub 2018 Jul 30. PMID 30061304
- [Background] Ma C, Li Z, Tong Y, Zhao M, Magnussen CG, Xi B. Leisure sedentary time and suicide risk among young adolescents: Data from 54 low- and middle-income countries. J Affect Disord. 2022 Feb 1;298(Pt A):457-463. doi: 10.1016/j.jad.2021.11.025. Epub 2021 Nov 12. PMID 34780860